CLINICAL TRIAL: NCT02514356
Title: A Small Randomized Controlled Trial Providing Weekly Information by SMS About Own and Group-level ARV Adherence to Patients in Two Clinics in Uganda
Brief Title: SMS as an Incentive To Adhere (SITA) - An Intervention Communicating Social Norms by SMS to Improve ARV Adherence
Acronym: SITA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: The AIDS Support Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R21MH107218-01 (NIH)
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: behavioral economics; antiretroviral adherence; SMS; mobile health (mHealth); Adolescents; Uganda; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Own adherence (Active Comparator): Participants in this group receive a weekly message by SMS. They receive the intervention 'Behavioral: Own Adherence'.
  Interventions: Behavioral: Own adherence
- Own and group level adherence (Active Comparator): Participants in this group receive a weekly message by SMS. They receive the intervention 'Behavioral: Own and Group Adherence'.
  Interventions: Behavioral: Own and group level adherence

INTERVENTIONS:
Behavioral: Own adherence — In this intervention group, participants receive weekly SMS messages informing them of their adherence that week as measured by the wise pill device used by the participant.
  Arms: Own adherence
Behavioral: Own and group level adherence — In this intervention group, participants receive weekly SMS messages informing them of their adherence that week as measured by the wise pill device used by the participant. In addition, in the same message they are informed of the adherence demonstrated by the other participants
  Arms: Own and group level adherence

SUMMARY:
The purpose of this study 'SMS as an Incentive To Adhere' (SITA) is to test two novel approaches of using SMS messages (provision of information about electronically measured own adherence, as well as in combination with group adherence level) to improve adherence to anitretroviral (ART) and pre-ART prophylaxis among youth age 15-24 at an HIV clinic in Uganda.

DETAILED DESCRIPTION:
SITA addresses two behavioral biases observed in people living with HIV/AIDS (PLWHA). The growing field of behavioral economics (BE) suggests that people display behavioral biases (i.e. systematic decision making errors) that among patients can contribute to suboptimal adherence. Investigators observed two important such biases in our own work in Uganda: first, investigators found that patients to a large degree overestimate their own adherence, i.e. think that they adhere better than they actually do. Second, a patient's social environment matters: PLWHA clearly care about their peers and their peers' attitudes and behavior.

SITA is based on Social Cognitive Theory (SCT) and adapts two traditional interventions to mHealth. The first intervention is that of self-monitoring, i.e. providing participants with feedback about their adherence performance. Traditionally this involves clinic visits that take up provider and patient time and resources; SITA instead suggests providing objective, real-time information measured by electronic monitoring (Wisepill) devices sent to patients by weekly SMS. Such feedback builds self-efficacy, a key SCT concept and thereby may improve adherence. The second intervention is based on the SCT concept of social learning. Perceived group norms, and interventions that affect those perceptions, are a key influence on health behavior among youths, providing a substitute for direct learning. Investigators adapt this approach to a mHealth environment by providing PLWHA not only with their own adherence information but also that of a reference (peer) group.

SITA will use mixed methods research techniques and focus on knowledge transfer within a multidisciplinary team. In formative Phase 1 investigators will conduct qualitative focus groups with key stakeholders to elicit information about the use of wisepill devices, and acceptance, feasibility and locally appropriate adaptation of SITA. In Phase 2, investigators will implement a nine-months, three-arm (with 50-60 participants each) randomized controlled trial: youths in intervention group 1 will receive information about their wisepill-measured adherence level by weekly SMS. Intervention group 2 will in addition be sent the adherence level of a reference group that investigators hypothesize to exert normative influence. The control group will receive the usual standard of care. Throughout the study investigators will focus on capacity building and knowledge transfer to the Ugandan collaborators through workshops and mentoring.

ELIGIBILITY:
Inclusion Criteria:

* have been in HIV care at the clinic for at least three months
* are currently taking HIV-related medication (ART or co-trimoxazole)
* either own a phone or have regular access to one
* intend to stay at the clinic for the study period
* are not in boarding school (where phones are forbidden)

Exclusion Criteria:

* does not speak or understand either English or Luganda
* does not have the cognitive capacity to consent and/or understand the study procedures

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 147 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Medication adherence rates using electronically monitored adherence (wise pill) data | 9 months after enrollment
  Wisepill data will be collected continuously over the course of the 9-month study period (preceded by about one month of adherence measurement only to allow for solution of any wisepill-related problems) allowing us to investigate daily adherence and its timing. Wisepill data indicating the date and time when the participant opened their pill container (either one of the ART medications or prophylaxis if not on ART yet) will be used to calculate the primary outcome variable of adherence (# of actual bottle openings / # of prescribed bottle openings).

SECONDARY OUTCOMES:
Self-reported adherence | 9 months after enrollment
  Survey will ask about self-reported adherence at baseline and month 9.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Linnemayr, PhD, Principal Investigator — RAND
Locations (1):
- The Aids Support Organization, Kampala, Uganda

REFERENCES:
- [Derived] MacCarthy S, Wagner Z, Mendoza-Graf A, Gutierrez CI, Samba C, Birungi J, Okoboi S, Linnemayr S. A randomized controlled trial study of the acceptability, feasibility, and preliminary impact of SITA (SMS as an Incentive To Adhere): a mobile technology-based intervention informed by behavioral economics to improve ART adherence among youth in Uganda. BMC Infect Dis. 2020 Feb 24;20(1):173. doi: 10.1186/s12879-020-4896-0. PMID 32093630
- [Derived] MacCarthy S, Saya U, Samba C, Birungi J, Okoboi S, Linnemayr S. "How am I going to live?": exploring barriers to ART adherence among adolescents and young adults living with HIV in Uganda. BMC Public Health. 2018 Oct 4;18(1):1158. doi: 10.1186/s12889-018-6048-7. PMID 30286746